CLINICAL TRIAL: NCT00050830
Title: A Phase 2, Randomized, Open-Label Study Of Single Agent CI-1033 In Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4161003
Record Dates: First submitted 2002-12-20; First posted 2002-12-24 (Estimated); Last update posted 2006-11-08 (Estimated); Status verified 2006-01

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Canertinib

INTERVENTIONS:
Drug: CI 1033

SUMMARY:
The purpose of study to determine the activity of CI 1033 against tumors in patients with advanced or metastatic NSCLC who have failed prior platinum-based combination chemotherapy. Another objective is to determine the safety of CI 1033.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented diagnosis of progressive or recurrent, locally advanced or metastatic NSCLC; a tumor that expresses at least one member of the erbB family of receptors; failed or relapsed after receiving a platinum-containing regimen as therapy; at least one measurable target lesion as defined by RECIST that has not been irradiated.

Exclusion Criteria:

* Prior exposure to agents that target the erbB receptor family; unknown response to prior platinum-containing chemotherapy regimen; cytotoxic chemotherapy within 3 weeks prior to baseline disease assessments (6 weeks for nitrosoureas or mitomycin); more than 2 prior chemotherapy regimens: immunotherapy or other biologic therapy within 2 weeks prior to baseline disease assessment; prior irradiation to areas encompassing greater than 30% of marrow-bearing bone; brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163
Dates: Start 2003-01; Study Completion 2005-11

PRIMARY OUTCOMES:
The primary objective is to assess the antitumor activity of CI 1033 in patients with advanced (progressive or recurrent, locally advanced [TNM Stage IIIB] or metastatic [TNM Stage IV]) NSCLC who have failed prior platinum-based combination chemotherapy

SECONDARY OUTCOMES:
Secondary objectives also include determining the safety of CI 1033 and the detection of any correlations between baseline tumor erbB expression and efficacy. Safety will be assessed by spontaneous AE reporting, physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- United States (33):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Greenbrae, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, San Mateo, California
  - Pfizer Investigational Site, San Pablo, California
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Park Ridge, Illinois
  - Pfizer Investigational Site, Skokie, Illinois
  - Pfizer Investigational Site, Jefferson, Indiana
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, La Grange, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Chippewa Falls, Wisconsin
  - Pfizer Investigational Site, Eau Claire, Wisconsin
  - Pfizer Investigational Site, Ladysmith, Wisconsin
  - Pfizer Investigational Site, Marshfield, Wisconsin
  - Pfizer Investigational Site, Minocqua, Wisconsin
  - Pfizer Investigational Site, Rice Lake, Wisconsin
  - Pfizer Investigational Site, Stevens Point, Wisconsin
  - Pfizer Investigational Site, Wausau, Wisconsin
  - Pfizer Investigational Site, Wisconsin Rapids, Wisconsin
  - Pfizer Investigational Site, Woodruff, Wisconsin
- Canada (2):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Montreal, Quebec
- Germany (3):
  - Pfizer Investigational Site, Gauting
  - Pfizer Investigational Site, Großhansdorf
  - Pfizer Investigational Site, Heidelberg
- Ireland (2):
  - Pfizer Investigational Site, Cork
  - Pfizer Investigational Site, Dublin
- Italy (2):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Orbassano (Torino)
- Pfizer Investigational Site, Amsterdam, North Holland, Netherlands
- Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona, Spain
- United Kingdom (2):
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, London